CLINICAL TRIAL: NCT04877405
Title: Retrospective Study to Identify Correlations Between the Clinical Parameters, Analytics and Neuroimaging Data in Patients That Suffered of Intraparenchymal Cerebral Hemorrhage
Brief Title: Retrospective Study of Intracerebral Hemorrhage Patients in Hospital Parc Taulí
Status: Completed | Type: Observational
Sponsor: Universitat Autonoma de Barcelona (Other)
Collaborators: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Santiago Rojas Codina MD PhD, Principal investigator, Universitat Autonoma de Barcelona
Other Study IDs: UHA-2021-1
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracerebral hemorraghe: Patients that suffered an intracerebral hemorraghe and that have been subjected to CT and MRI scans
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This observational study is not focused on therapeutic intervention

SUMMARY:
This is a retrospective observational study to investigate the clinical, analytical and neuroimaging data generated during routine clinical management of intracerebral hemorrhage. The study will review the data from about 500 patients attended during the last ten years in the Neurology Department of Hospital Parc Taulí de Sabadell.

The aim is to measure the size of the lesion in neuroimage (TC and MRI), the edema, the alterations in diffusion weighted images and to correlate this data with clinical parameters and analytical measurements. With this approach investigators plan to investigate the incidence of hematoma growth, the role of perilesional edema and diffusion changes, and the relation between neuroimaging findings and clinical outcome. The study also try to establish significant correlations between clinical and analytical data, the clinical outcome and and the magnitude of changes in neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been attended at the Hospital Parc Taulí for the last 10 years after presenting an intraparenchymal hemorrhage.
* The patients have had to undergo a computed tomography at the admission and a cranial magnetic resonance during the hospitalization in the time course specified in point in the protocol
* The patients must present in their clinical story the analytical determinations detailed in the protocol.

Exclusion Criteria:

* Intracerebral hemorrhage secondary to head trauma
* Intracerebral hemorrhage secondary to neoplasm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consist in the patients attended due to spontaneous intracerebral hemorrhage in Hospital Parc Taulí de Sabadell during the last decade. Traumatic or oncologic origin of the hemorrhage constitute exclusion criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Hematoma growth | 2 days
  Difference of hematoma size between CT conducted at admission and MRI conducted during follow up
Correlation between hematoma growth and clinical paramenters | 2 days
  Determine the clinical parameters related with hematoma growth
Correlation between hematoma growth and analytical parameters | 2 days
  Determine the analytical parameters related with hematoma growth
Perilesional edema | 2 days
  Size of edema measured in FLAIR sequences
Correlation between clinical parameters and the size of edema measured in FLAIR sequences | 2 days
  Determine the relationship between clinical parameters and the size of edema
Correlation between analytical parameters and the size of edema measured in FLAIR sequences | 2 days
  Determine the relationship between analytical parameters and the size of edema
Alterations in DWI | 2 days
  Size of alterations in diffusion weighted image
Correlation between clinical parameters and the size of alterations in DWI | 2 days
  Determine the relationship between clinical parameters and the size of alterations in DWI
Correlation between analytical parameters and the size of alterations in DWI | 2 days
  Determine the relationship between analytical parameters and the size of alterations in DWI
Correlation between hematoma growth and clinical outcome | 1 month
  Determine the impact of hematoma growth on clinical outcome
Correlation between perilesional edema size and clinical outcome | 1 month
  Determine the relationship between the size of edema and clinical outcome
Correlation between the size of DWI alterations and clinical outcome | 1 month
  Determine the relationship between the size of DWI alterations and clinical outcome
Correlation between the clinical parameters and clinical outcome | 1 month
  Determine the relationship between the clinical parametes and clinical outcome
Correlation between the analyticial parameters and clinical outcome | 1 month
  Determine the relationship between the analytical parametes and clinical outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Santiago Rojas Codina MD PhD, Cerdanyola del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared with other researchers under request